CLINICAL TRIAL: NCT04425837
Title: Effectiveness and Safety of Convalescent Plasma in Patients With High-risk COVID-19: A Randomized, Controlled Study CRI-CP (Coronavirus Investigation - Convalescent Plasma)
Brief Title: Effectiveness and Safety of Convalescent Plasma in Patients With High-risk COVID-19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundación Santa Fe de Bogota (Other)
Responsible Party: Principal Investigator, Guillermo Enrique Quintero-Vega, Hematologist, Fundación Santa Fe de Bogota
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PLASMA COVID-19
Record Dates: First submitted 2020-05-29; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Sars-CoV2; Covid-19
Keywords: COVID-19 serotherapy; Mortality; Safety
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Serotherapy; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care alone (Active Comparator)
  Interventions: Other: Standard care
- SARS-CoV-2 convalescent plasma treatment plus standard care (Experimental)
  Interventions: Biological: SARS-CoV-2 convalescent plasma treatment; Other: Standard care

INTERVENTIONS:
Biological: SARS-CoV-2 convalescent plasma treatment — Plasma transfusion of convalescent patients from COVID-19 with negative RT-PCR, and antibody titers of 1:160 or greater at a dose of 400ml distributed in two doses administered on the same day intravenous administration
  Arms: SARS-CoV-2 convalescent plasma treatment plus standard care
Other: Standard care — Standard care according to guidelines and national regulations

SUMMARY:
The severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) has affected the global population with significant morbidity and mortality. One of the main concerns is the management of the patients since there is no specific treatment for this condition. Therefore, in SARS-CoV-2 patients the compassionate use of off-label therapies has been initiated; such as the use of plasma from convalescent patients. This treatment has been used in other pandemics like SARS-CoV-1, H5N1, H1N1, Ebola, among others. This study is a phase II/III randomized clinical trial to assess the effectiveness and safety of convalescent plasma administration in patients with high-risk SARS-CoV-2.

DETAILED DESCRIPTION:
This is a Phase II/III randomized clinical trial to assess the effectiveness and safety of anti-SARS-CoV-2 convalescent plasma in i) hospitalized adult patients with high-risk of progression SARS-CoV-2 infection and ii) patients in Intensive Care Unit (ICU).

Compatible ABO plasma from convalescent patients will be administered at a dose of 400 ml divided into two doses intravenously. Outcomes will be measured as follows:

* Group of patients with critical illness:

Primary outcomes (Effectiveness and safety):

* Mortality
* Safety: Presence of adverse events

Secondary outcomes:

* Intensive care unit length of stay
* Evolution of clinical and paraclinical aspects.

  * Group of patients at high risk of progression:

Primary outcomes (Effectiveness and safety):

* Mortality
* Safety: Presence of adverse events
* Admission to ICU in 30 days
* Mechanical ventilation requirement

Secondary outcomes:

* Hospital/Intensive care unit length of stay
* Evolution of clinical and paraclinical aspects.

ELIGIBILITY:
Inclusion Criteria:

All patients

* Patients diagnosed with COVID-19 infection by RT-PCR technique
* Patients ≥ 18 years of age
* Patients in standard care according to the national guide
* Onset of symptoms ≤ 14 days
* Signature of informed consent report

Patients at high risk of progression, defined by all of the following:

* Score greater than 9 on the CALL scale
* Pao2 / Fio2 ≤ 200 (parameters adjusted to the height of Bogotá, Colombia)
* X-ray or CT compatible with pneumonia
* Hospitalized patients

Critically ill patients, defined by any of the following:

* Mechanical ventilation requeriment
* Patients in Intensive Care Unit or Intermediate Care Unit
* Ventilatory failure, septic shock, dysfunction or multi-organ failure

Exclusion Criteria:

* Negative RT-PCR result from secretion 48 hours prior to study recruitment
* History of allergic reaction to blood or plasma in patients with a known history of IgA deficiency
* Patients participating in other clinical trial
* History of allergy to blood products
* History of confirmed infection and that required antibiotic or antifungal treatment 30 days prior to recruitment
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Mortality | Up to 30 days after the study enrollment
  Death of the patient (yes/no)
Adverse events | Up to 30 days after the study enrollment
  Presence of any of the following adverse events (yes/no):
  1. Nonhemolytic febrile reactions
  2. Allergic reactions
  3. Acute hemolytic reactions
  4. Non-immune hemolysis
  5. Acute transfusion-related lung damage
  6. Transfusion-related circulatory overload
  7. Metabolic reactions
  8. Hypotensive reactions
  9. Delayed hemolytic reactions
  10. Post transfusion purple
  11. Graft versus host disease
  12. Bacterial contamination of blood components
  13. Viral infections
  14. Other infections (syphilis, prions, malaria, Chagas, yellow fever, dengue)
ICU admission | Up to 30 days after the study enrollment
  Admitted to intensive care units (ICUs) (yes/no)
Mechanical ventilation | Up to 30 days after the study enrollment
  Mechanical ventilation requirement (yes/no)

SECONDARY OUTCOMES:
ICU length | Up to 30 days after the study enrollment
  Intensive care unit length of stay
Reduction of D Dimer | Assessment at day 30 after study enrollment
  D dimer reduction below 1mcg / ml
LDH reduction | Assessment at day 30 after study enrollment
  Reduction of LDH below 350 IU / L
Reduction of Troponin level | Assessment at day 30 after study enrollment
  Reduction of troponin level to than 8 pg / mL
Decrease in ferritin level | Assessment at day 30 after study enrollment
  Decrease in ferritin level below 1025 mcg / L
Decrease in procalcitonin level | Assessment at day 30 after study enrollment
  Decrease in procalcitonin level below 0.1ng / ml
Decrease in CRP | Assessment at day 30 after study enrollment
  Decrease in CRP level bellow <8 mg / L
Increase in lymphocyte count | Assessment at day 30 after study enrollment
  Increase in lymphocyte count greater than 0.6 x 10-9 / L
Increase in PaO2 / Fio2 | Assessment at day 30 after study enrollment
  Increase in PaO2 / Fio2 greater than 200
Decrease in Sequential Organ failure assessment (SOFA ) score | Assessment at day 30 after study enrollment
  Scale of 24 points, greater number indicates worst outcome
Extracorporeal membrane oxygenation (ECMO) | Assessment at day 30 after study enrollment
  Extracorporeal membrane oxygenation requirement (ECMO)
Lung infiltration | Assessment at day 30 after study enrollment
  Decrease in the percentage of lung infiltration

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación Santa Fe de Bogotá, Bogotá, Cundinamarca, Colombia